CLINICAL TRIAL: NCT04484298
Title: Dynamic Variation of Impedance Cardiography (ICG) a Diagnostic Tool of Acute Heart Failure (AHF) in Emergency Department (ED) Patients Admitted for Acute Dyspnea
Brief Title: Dynamic Variation of Impedance Cardiography(DYVIC) as a Diagnostic Tool of Acute Heart Failure (AHF)
Acronym: dyvic2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, professor semir nouira, University of Monastir
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: DYVIC2
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Heart Failure
Keywords: dyspnea; acute; heart failure; bio-impedance; biopac system
MeSH Terms: conditions — Heart Failure; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reference group (Experimental): patients presenting to the emergency department with acute onset dyspnea are assessed for acute heart failure using the bio impedance technology (BIOPAC system) to measure the cardiac output in different clinical situations.
  FIRST: the cardiac output (CO) is measured at the reference position. Inbetween each step the patient was put in the reference position during 5 minutes.
  Interventions: Diagnostic Test: Reference position patient is put in a 30 degree supine position during 5 minutes
- TRINITRINE (Experimental): 0.6 mg of nitroglycerin was given to the patient sublingual and we measure the cardiac output by BIOPAC system(0.6 mg of Nitroglycerin was administered sublingually and CO was evaluated.
  Interventions: Diagnostic Test: nitroglucerin

INTERVENTIONS:
Diagnostic Test: Reference position patient is put in a 30 degree supine position during 5 minutes — Each patient is initially placed in a semi-sitting position at 30° for 5 minutes and then CO is measured (baseline CO)
  Arms: reference group
Diagnostic Test: nitroglucerin — 0.6 mg of Nitroglycerin was administered by sublingual root and CO was evaluated.
  Arms: TRINITRINE

SUMMARY:
the study aimed to evaluate the diagnostic performance of cardiac output (CO) change after the use of trinitrine in the diagnosis of heart failure patients with acute dyspnea.

DETAILED DESCRIPTION:
Acute heart failure (AHF) is a frequent condition in emergency department and is responsible of high number of admissions, complications, and deaths.

despite advances in diagnostic techniques, AHF diagnosis still be challenging .

Measurement of cardiac output (CO) is used to evaluate global cardiac function and changes in CO may be used to identify a change in the hemodynamic status of patient.

the gold standard of measuring CO is thermodilution catheterization, however it is an invasive technique with high risks.

Impedance cardiography (ICG) is a noninvasive method for measuring CO. it is performed by applying small electrical current to the chest through electrodes placed on the neck and sides.

the pulsatile flow of blood causes fluctuations in the current, and the device calculates CO from the impedance waveform.

In practice, the investigators connect the device "BIOPAC" by using four electrodes which the investigators place on the base of the neck (posterior face) and on the base of the thorax (posterior face).

The ECG recording is taken simultaneously with two other electrodes placed at the right upper limb and left lower limb.

In addition to detecting the electric current and the ECG, heart sounds are recorded using a sensor that is placed at the mitral site.

Each patient is initially placed in a semi-sitting position at 30° for 5 minutes and then CO is measured (baseline CO). NTG (0.6 mg) is then given to the patient sublingually and CO measurement was repeated. CO is calculated by averaging three measurements at one minute intervals at baseline and after NTG administration. DeltaCO was defined as the percent of change of baseline CO after NTG test.

ELIGIBILITY:
Inclusion Criteria:

* 18 year old or above non traumatic acute dyspnea

Exclusion Criteria:

* ECG diagnostic for acute myocardial infarction or ischemic chest pain within the prior 24 hours,
* pericardial effusion ,
* chest wall deformity suspected of causing dyspnea,
* coma,
* need for mechanical ventilation or vasopressor drugs,
* serious and sustained arrhythmia,
* pace maker,
* severe mitral valve disease, severe pulmonary arterial hypertension,
* renal failure (creatinine >350µmol/l.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Cardiac output variation measured by ICG before and after nitroglycerin in acute dyspneic patients between the AHF and non AHF groups | 24 hours
  the diagnostic performance is evaluated by calculating the CO in ml/min by bio-impedance technique and compare the values between patients with and without AHF and between baseline.
roc curve | 24
  Receiver operating characteristic (ROC) curves for predicting HF were constructed and area under curve (AUC) was measured for the deltaCO.
Sensitivity, specificity, positive and negative predictive values, and likelihood ratios of positive and negative results were calculated using the optimal cutoff value of deltaCO. | 24 hours
  Sensitivity, specificity, positive and negative predictive values, and likelihood ratios of positive and negative results were calculated using the optimal cutoff value of deltaCO.

CONTACTS AND LOCATIONS:
Overall Officials: nouira semir, MD, Principal Investigator — University of Monastir
Locations (1):
- Emergency department of fattouma bourguiba university hospital, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No